CLINICAL TRIAL: NCT05505903
Title: Influence of Duration Since Birth Until Admission to Well-baby Nursery on Neonatal Temperature at Admission
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Principal Investigator, Hillel Yaffe Medical Center
Other Study IDs: 0032-22-HYMC-IL
Record Dates: First submitted 2021-10-04; First posted 2022-08-18 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Hypothermia, Newborn
Keywords: hypothermia; friendly Cesarean section
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaginal delivery: Newborn Infants born by vaginal delivery.
  Interventions: Diagnostic Test: Temerature measurement
- Regular Cesarean section: Newborn infants born by regular Cesarean section
  Interventions: Diagnostic Test: Temerature measurement
- Friendly Cesarean section: Newborn infants born by friendly Cesarean section
  Interventions: Diagnostic Test: Temerature measurement

INTERVENTIONS:
Diagnostic Test: Temerature measurement — Temerature measurement on admission to WBN or NICU

SUMMARY:
The investigators will collect the time interval from birth to arrival to WBN or NICU, the time interval from arrival to nurse admission, the first measured temperature, and the week of birth.

The investigators will divide the newborn infants to three groups: infants born vaginally, infants born by regular Cesarean section, and infants born by friendly Cesarean section, and compare the groups.

DETAILED DESCRIPTION:
Introduction Friendly Cesarean section mimics normal vaginal delivery as the newborn is put on mother's chest immediately after delivery and cutting the umbilical cord, and the mother even breastfeeds the newborn infant, if she wishes to. Friendly Cesarean section is offered to the mother if there are no contraindications, such as general anesthesia, fetal distress, or prematurity. Skin to skin contacts lasts for several minutes, as long as the mothers wish to, and depend on mothers' medical state, and newborns' medical state.

In friendly Cesarean section, the skin to skin contact technique includes putting the newborn on mother's chest, and covering them both by a blanket. Yet, during Cesarean section the mother is covered by a thin paper-like sterile sheet, and as the temperature in operating room is low, her skin cools gradually from the spinal anesthesia until actually delivering the newborn infant. So, although the newborn infant is put on the mother's chest and covered by a blanket, there is a possibility for it to develop hypothermia.

Literature about this issue is rare, so the investigators conducted a study to check this possibility.

Methods In Hillel Yaffe medical center nurses measure infants temperature on admission to well-baby nursery (WBN) or neonatal intensive care unit (NICU). Admission is not always performed on arrival, due to other nurse-tasks, such as other newborn infants treatment, or breastfeeding education.

The most measureable piece of data that characterize friendly Cesarean section is the longer time interval from the birth until arrival to WBN or NICU.

Inclusion criteria: infants born within the time study interval. Exclusion criteria: infants born at less than complete 35 gestational weeks, since there is no for offer friendly Cesarean section for these births.

The investigators will collect the time interval from birth to arrival to WBN or NICU, the time interval from arrival to nurse admission, the first measured temperature, and the week of birth.

The investigators will divide the newborn infants to three groups: infants born vaginally, infants born by regular Cesarean section, and infants born by friendly Cesarean section, and compare the groups.

ELIGIBILITY:
Inclusion Criteria:

* all newborn infants

Exclusion Criteria:

* infants born after less than 35 complete gestational weeks

Max Age: 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants born at Hillel Yaffe meducal center
Sampling Method: Non-Probability Sample
Enrollment: 2412 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Temperature | 1 year
  The temperature upon admission to WBN or NICU

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Study Chair — Hille Yaffe medical center
Locations (1):
- Neonatal intensive care unit, Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No